CLINICAL TRIAL: NCT04211636
Title: Maladaptive Systemic Immune Response After Spinal Cord Injury: Humoral Post-traumatic Autoimmunity Against Central and Peripheral Nervous System Antigens in Association With Neurogenous Immune Depression as a Confounder of Rehabilitation
Brief Title: Autoimmunity And Immune Deficiency After Spinal Cord Injury: Association With Rehabilitation Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Marcel Kopp, MD (Other)
Collaborators: Foundation Wings For Life (Other); University Hospital Tuebingen (Other); Unfallkrankenhaus Berlin (Other); Balgrist University Hospital (Other); I.R.C.C.S. Fondazione Santa Lucia (Other); University of Zurich (Other); Medical University of Vienna (Other); Ruhr University of Bochum (Other); Swiss Federal Institute of Technology (Other); King's College London (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Marcel Kopp, MD, Study Coordinator, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: SCIentinel-prolong
Record Dates: First submitted 2019-12-20; First posted 2019-12-26 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Spinal Cord Trauma
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, peripheral blood mononuclear cells, cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Complete SCI, AIS A: Patients with complete spinal cord injury (AIS A)
- Incomplete SCI, AIS B, C, D: Patients with incomplete spinal cord injury (AIS B, C, D)
- Vertebral injuries without SCI: Patients with vertebral injuries without spinal cord injury (control)

SUMMARY:
The SCIentinel-prolong study systematically analyzes humoral autoantibody responses and thier interaction with post-spinal cord injury (SCI) immune-deficiency and infections as well as their association with the clinical course of rehabilitation. Therefore, molecular and immunological tests in blood and cerebrospinal fluid specimen are combined with clinical outcomes ranging from neurological function, neuropathic pain and spasticity to walking tests and measures of independence in daily living within the first year after SCI. Including a control group with participants suffering from vertebral fractures without SCI allows to differentiate between neurological and general injury and treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Acute traumatic SCI, American Spinal Injury Association Impairment Scale (AIS) A to D, neurologic level of injury C3 - L2 or acute vertebral fracture without SCI
* Inclusion within 21 days post-injury
* For Italian centers only: SCI-Treatment using Methylprednisolone (according to NASCIS).

Exclusion Criteria:

* Non-traumatic SCI
* Severe multiple trauma
* Serious traumatic brain injury
* Pre-exiting neurological diseases
* Malignant Neoplasia, except in complete remission for 5 years
* Rheumatic diseases / collagenosis / vasculitis
* Other autoimmune diseases
* Pre-existing chronic infection
* Severe alcohol or drug addiction
* Pregnancy or lactation
* Simultaneous participation in interventional clinical trials
* For centers in Germany or Switzerland only: SCI-treatment using Methylprednisolone (according to NASCIS).

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants from primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic autoimmunity | 3 months (10-14 weeks) post injury
  Prevalence of autoantibodies against central and peripheral nervous system antigens in cerebrospinal fluid and serum

SECONDARY OUTCOMES:
International Standards for Neurological Classification of SCI - Upper Extremity Motor Score | 2 weeks, 3-6 weeks, 3 month, 6month, 1 year post injury
  Minimum 0, maximum 50; higher scores mean a better outcome
International Standards for Neurological Classification of SCI - Lower Extremity Motor Score | 2 weeks, 3-6 weeks, 3 month, 6month, 1 year post injury
  Minimum 0, maximum 50; higher scores mean a better outcome
International Standards for Neurological Classification of SCI - Sensory light touch score | 2 weeks, 3-6 weeks, 3 month, 6month, 1 year post injury
  Minimum 0, maximum 112; higher scores mean a better outcome
International Standards for Neurological Classification of SCI - Sensory pin prick score | 2 weeks, 3-6 weeks, 3 month, 6month, 1 year post injury
  Minimum 0, maximum 112; higher scores mean a better outcome
American Spinal Injury Association Impairment Scale | 2 weeks, 3-6 weeks, 3 month, 6month, 1 year post injury
  Ordinal alphabetical scale. Range A to E. Change in the scale to one of the subsequent letters in the alphabet means a better outcome.
Spinal Cord Independence Measure III | 2 weeks, 3-6 weeks, 3 month, 6month, 1 year post injury
  Composite instrument for the assessment of physical independence; minimum 0, maximum 100; higher scores mean a better outcome
Walking Index for Spinal Cord Injury II | 2 weeks, 3-6 weeks, 3 month, 6month, 1 year post injury
  Score for walking ability; minimum 0, maximum 20; higher scores mean a better outcome
10m-walk-test | 2 weeks, 3-6 weeks, 3 month, 6month, 1 year post injury
  Time in seconds required for 10 meter walking; higher scores mean a worse outcome
Timed-up-and go | 2 weeks, 3-6 weeks, 3 month, 6month, 1 year post injury
  Time in seconds needed to raise from a chair, walk a distance of 3 m, turn back and sit down again; higher scores mean a worse outcome
6-minutes-walk-test | 2 weeks, 3-6 weeks, 3 month, 6month, 1 year post injury
  Walking distance in meters covered in 6 minutes; higher scores mean a better outcome
Neuropathic Pain Scale 10 | 2 weeks, 3-6 weeks, 3 month, 6month, 1 year post injury
  Instrument comprising 10 numeric analogue scales for intensity and qualities of pain; each item ranges from 0-10; higher scores mean a worse outcome
Spinal Cord Injury Pain Basic Dataset | 2 weeks, 3-6 weeks, 3 month, 6month, 1 year post injury
  Composite instrument for the assessment of pain locations, type and intensity
Modified Ashworth Scale | 2 weeks, 3-6 weeks, 3 month, 6month, 1 year post injury
  Assessment of muscle tone and resistance to passive motion; minimum 0, maximum 4, higher scores mean a worse outcome
Penn spasm frequency scale | 2 weeks, 3-6 weeks, 3 month, 6month, 1 year post injury
  Patient rated frequency of spasms; minimum 0, maximum 4; higher scores mean a worse outcome
Somatosensory evoked potentials | 2 weeks, 3 months
  Tibial nerve and ulnar nerve; response is graded as ranging from 1=abolished to 4=normal response; higher scores mean better outcome
Motor evoked potentials | 2 weeks, 3 months
  Anterior tibial muscle, abductor hallucis, abductor digiti minimi; response is graded as ranging from 1=abolished to 4=normal response; higher scores mean better outcome
Electroneurography | 2 weeks, 3 months
  Abductor hallucis and abductor digiti minimi; latency, amplitude and F-waves
Sympathetic skin response | 2 weeks, 3 months
  Skin response at palm and sole
Human Leukocyte Antigen - DR isotype expression on monocytes | 1 day, 3 days, 1week, 2 weeks, 3-6 weeks, 3 months, 6 months, 1 year post injury
  Anti-Human Leukocyte Antigen - DR isotype antibodies bound per monocyte, higher values mean better outcome
Immune phenotyping | 1 day, 3 days, 1week, 2 weeks, 3-6 weeks, 3 months, 6 months, 1 year post injury
  Panel of T-lymphocyte and B-lymphocyte subpopulations
Functional immune assays | 1 day, 3 days, 1week, 2 weeks, 3-6 weeks, 3 months, 6 months, 1 year post injury
  White blood cell ex-vivo stimulation
Damage Associated Molecular Patterns | 1week, 3 months,
  Immunoassays in plasma and CSF
Markers of Ferroptosis | 1week, 3 months
  Immunoassays in plasma and CSF

CONTACTS AND LOCATIONS:
Overall Officials: Jan M Schwab, MD, PhD, Study Chair — Ohio State University; Marcel A Kopp, MD, Study Director — Charite University, Berlin, Germany